CLINICAL TRIAL: NCT06841705
Title: Early Concomitant Vedolizumab as First-Line for Immune-Related Colitis Therapy Trial
Brief Title: Early Vedolizumab as First-Line for Immune-Related Colitis Therapy Trial
Acronym: EVITA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shilpa Grover, MD, MPH (Other)
Collaborators: Dana-Farber/Brigham and Women's Cancer Center (Other); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Shilpa Grover, MD, MPH, Director Onco-Gastroenterology, Division of Gastroenterology, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-080
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Immune Checkpoint Inhibitor-Related Colitis
Keywords: Immunotherapy Colitis; Immune Checkpoint Inhibitor Colitis; ICI Colitis; Colitis
MeSH Terms: conditions — Colitis | interventions — vedolizumab; Injections; Prednisone; Methylprednisolone; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vedolizumab and Short Course of Steroids (Experimental): Participants in this arm will receive Vedolizumab infusions (3 doses) and steroids for 10 days (intravenous Medrol daily for 3 days and Prednisone daily for 7 days). Participants may also receive daily placebo (for Prednisone and Sulfamethoxazole-Trimethoprim).
  Interventions: Drug: Vedolizumab 300 MG Injection [Entyvio]; Drug: Prednisone (and methylprednisolone); Other: Placebo Prednisone Capsules; Drug: Placebo for Sulfamethoxazole-Trimethoprim
- Standard Course of Steroids (Active Comparator): Participants in this arm will receive steroids for 10 days (intravenous Medrol daily for 3 days and Prednisone daily for 7 days), followed by a steroid (Prednisone) taper. Participants may also receive Sulfamethoxazole-Trimethoprim (an antibiotic). Participants will receive 3 placebo infusions.
  Interventions: Drug: Prednisone (and methylprednisolone); Drug: Prednisone Taper; Other: Placebo Vedolizumab; Other: Sulfamethoxazole-Trimethoprim

INTERVENTIONS:
Drug: Vedolizumab 300 MG Injection [Entyvio] — This is a biologic medication to treat colitis
  Other Names: Entyvio
  Arms: Vedolizumab and Short Course of Steroids
Drug: Prednisone (and methylprednisolone) — This is a steroid
Drug: Prednisone Taper — This is a tapering dose of prednisone
  Arms: Standard Course of Steroids
Other: Placebo Prednisone Capsules — Placebo for Prednisone
  Arms: Vedolizumab and Short Course of Steroids
Other: Placebo Vedolizumab — Placebo for Vedolizumab
  Arms: Standard Course of Steroids
Other: Sulfamethoxazole-Trimethoprim — Antibiotic if on >21 days of steroids
  Arms: Standard Course of Steroids
Drug: Placebo for Sulfamethoxazole-Trimethoprim — Placebo for antibiotic (Sulfamethoxazole-Trimethoprim) Antibiotic. Only if on >21 days of prednisone/placebo
  Arms: Vedolizumab and Short Course of Steroids

SUMMARY:
The goal of this clinical trial is to compare the effectiveness and safety of Vedolizumab with a short course of steroids compared to standard course of steroids for the treatment of immune checkpoint inhibitor colitis (ICI colitis) in adults.

The main questions it aims to answer are:

* How many patients treated with Vedolizumab and a short course of steroids experience resolution of colitis at 8 weeks.
* How many patients treated with a standard course of steroids experience resolution of colitis at 8 weeks.

Participants will:

Recieve 3 doses of Vedolizumab or a placebo (a look-alike substance that contains no drug) infusions over 6 weeks Receive intravenous Medrol daily for 3 days Receive Prednisone daily for 7 days Receive Prednisone or placebo taper daily Receive Sulfamethoxazole-Trimethoprim or placebo taper daily Weekly checkups and periodic tests

DETAILED DESCRIPTION:
This is a phase II, randomized trial to evaluate the efficacy and safety of the drugs Vedolizumab, methylprednisolone, and prednisone to manage the side of effect of colitis caused by immune checkpoint inhibitors (ICIs).

The names of the treatments involved in this study are:

* Vedolizumab
* Methylprednisolone
* Prednisone
* Sulfamethoxazole-Trimethoprim

The FDA has approved Vedolizumab, methylprednisolone, and prednisone to treat many conditions affecting the immune system, including colitis.

Participants who enroll in this study will undergo one or more flexible sigmoidoscopies or colonoscopies as part of their clinical care. The first of these procedures would occur at the time of study enrollment, and the second may occur after several weeks of treatment at the discretion of the study doctor. During these procedures, biopsies will be collected for clinical purposes as well as for research purposes. Blood and stool samples will also be collected for research. Any extra samples for research would only be collected only if it is safe for the participant.

Participants will complete weekly follow-ups either over the phone or in-person. During these visits, participants will be asked about any new symptoms or changes in their health, their medications, and their symptoms. Blood for research may be collected at four of these visits if it coincides with a scheduled clinical blood draw.

Participants are expected to be on study treatment for 8 weeks. The study team will review their medical records at 12 months for any changes in their health.

It is expected that approximately 80 people will participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* In order to participate in the study, a patient must meet all the following inclusion criteria:
* Age ≥18 years.
* Treatment with an ICI for cancer within the past 8 weeks.
* Confirmed endoscopic/histologic diagnosis of ICI colitis.
* Grade 2-3 diarrhea by Common Terminology Criteria for Adverse Events.
* Willing and able to comply with the requirements of the protocol.
* Ability to understand and the willingness to sign a written informed consent document.
* Exclusion Criteria
* Prior history of inflammatory colitis requiring treatment with greater than prednisone 10 mg daily or equivalent or any immunosuppressive medication.
* Current or recent use of immunosuppressive biologic medication (for any reason including ICI colitis) within 4 weeks.
* Concurrent immune-related adverse event requiring systemic steroids or systemic immunosuppression within 2 weeks.
* Colonic perforation or abscess.
* Partial or complete bowel obstruction within the last 3 months, signs/symptoms of bowel obstruction, or known radiologic evidence of impending obstruction.
* Active Clostridium difficile or other colonic infection.
* Concurrent hepatitis B or C infection.
* History of untreated tuberculosis and/or positive quantiferon/Tspot test without previous tuberculosis prophylaxis, or untreated active infection with mycobacterium tuberculosis.
* Active or known prior infection with nontuberculous mycobacteria (NTM).
* Unable or unwilling to undergo a colonoscopy/flexible sigmoidoscopy.
* Inpatient status, though patients can be screened while inpatients, they must be outpatient for the planned treatment of ICI colitis.
* History of total proctocolectomy.
* Female patients who are pregnant or breastfeeding or plan to become pregnant in the next 6 months.
* Patients who are unable to give informed consent.
* Previous SARS-CoV-2 infection within 10 days for mild infections or 20 days for severe/critical illness prior to first Vedolizumab dose.
* Unable to adhere to protocol requirements.
* Any condition that the physician investigators deem unsafe, including other conditions or medications that the investigator determines will put the subject at greater risk from vedolizumab plus brief course of steroids.
* Allergy to sulfamethoxazole-trimethoprim.
* Weight greater than 120 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Steroid-free remission rate | 8 weeks
  Defined as less than 10 mg of prednisone/day and grade 1 or lower diarrhea symptoms without the use of additional biologic rescue medication.

SECONDARY OUTCOMES:
Steroid-free remission rate | 5 weeks
  Defined as less than 10 mg of prednisone/day and grade 1 or lower diarrhea symptoms without the use of additional biologic rescue medication.
Change in calprotectin | 0, 2, 5 and 8 weeks
  As compared to baseline
Cumulative steroid exposure | 5 weeks and 8 weeks
  Steroid dose x Duration of treatment
Time to steroid-free colitis remission | Up to 12 months
  Defined as the time from the first day of treatment to the first day with less than 10 mg of prednisone/day and grade 1 or lower symptoms.
Rate of secondary immunosuppression for management of ICI colitis | 5 weeks and 8 weeks
  Defined as the use of open-label prednisone or biologic rescue medication
Rate of symptomatic remission | 5 weeks and 8 weeks
  Defined as a reduction in stool frequency to < 4 bowel movements/day at 1 week
Hospitalization rate | 8 weeks
  Due to colitis
Rates of colectomy | 8 weeks
  Due to colitis
Endoscopic resolution of colitis | 8 weeks
  Rate of endoscopic resolution of colitis will be determined, if endoscopy is performed at 8 weeks
Best overall cancer response | 8 weeks and 12 months
Overall survival | Time of death or 12 months
  Defined as time from the first day of protocol treatment to death or last contact date.
Proportion of participants with an adverse event (AE) | 5 weeks
  Proportion of participants with an AE through week 5 (±5 days) attributable to ICI colitis treatment
Proportion of participants with an AE | 8 weeks
  Proportion of participants with an AE through week 8 (±5 days) attributable to ICI colitis treatment
Presence of histologic inflammation | 0, 8 weeks
Pattern of histologic inflammation | 0, 8 weeks
  Categorized as: Active Colitis Pattern, Lymphocytic Pattern, Graft Vs Host Disease Pattern, Mixed Pattern.

OTHER OUTCOMES:
Time to resumption of cancer treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Grover, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset that underlie results in a publication will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication. Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
Access Criteria: De-identified participant data from the final research dataset used in the published manuscript may be shared under the terms of a Data Use Agreement. Requests may be directed to sgrover@bwh.harvard.edu
  The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.